CLINICAL TRIAL: NCT04307069
Title: Comparison Between Two Protocols for Management of Prelabor Rupture of the Membranes at Term
Brief Title: Management of Prelabor Rupture of the Membranes at Term
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rambam Health-Care Center
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Fetal Infection; Chorioamnionitis; Endometritis; Cesarean Section Complications
MeSH Terms: conditions — Chorioamnionitis; Endometritis | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate oxytocin infusion (Experimental): Once the patient will arrive at the maternity ward with prelabor rupture of membranes, she will receive oxytocin for augmentation of labor.
  Interventions: Drug: Oxytocin
- Expectant management for 24 hours (Experimental): Once the patient will arrive at the maternity ward with prelabor rupture of membranes, we will wait for spontaneous delivery to occur. After 24 hours of rupture of membranes, the woman will receive oxytocin for augmentation of labor.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — The drug wil be adminisrate for augmentation of labor at admission.
  Other Names: pitocin

SUMMARY:
Prolonged rupture of membranes has been associated with increased risk of chorioamnionitis and endometritis. In this study the investigators will investigate whether an early intervention to augment labor with oxytocin is superior to expected management for spontaneous delivery (up to 24 hours).

DETAILED DESCRIPTION:
Prelabor rupture of the membranes (PROM) refers to rupture of the fetal membranes prior to the onset of regular uterine contractions.

PROM at term can be managed actively by induction of labor or expectantly by waiting for the onset of a spontaneous labor. Several studies have shown an association between expectant management and higher rates of maternal and neonatal adverse outcomes, especially infections. Furthermore, expectant management has been shown to increase the risk for cesarean deliveries (CD), chronic lung disease, cerebral palsy and neonatal mortality. It is suggested that the risk for those complications increase proportionally with the longer the duration of ruptured membranes. Others disagree with those associations.

In this study the investigators will investigate whether early administration of oxytocin is superior to expectant management of 24 hours in patients with PROM at term, in terms of time to delivery and maternal and neonatal adverse outcomes, regardless of bishop score.

ELIGIBILITY:
Inclusion Criteria:

1. Primiparous women with a singleton pregnancy that are admitted with prelabor rupture of membranes.
2. Women at gestational age 370/7 or more.
3. Vertex presentation.

Exclusion Criteria:

1. Age 18 and under.
2. High order gestation.
3. Women with contraindication for a vaginal delivery.
4. Active labor.
5. Documented fetal anomalies.
6. Known or suspected intrauterine infection (temperature > 38 degrees, leucocytosis).
7. Non reassuring fetal heart rate tracing.
8. Positive group B streptococcus status.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 524 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Maternal infectious morbidity | Up to 48 hours postpartum
  Maternal chorioamnionitis and/ or endometritis

SECONDARY OUTCOMES:
Length of latent and active phases of labor. | During Labor
  According to vaginal examinations during labor
Adverse maternal outcome | Up to 48 hours postpartum
  infectious (chorioamnionitis/endometritis), serious maternal morbidity and mortality (death, cardiac arrest, respiratory arrest, ICU admission), post-partum hemorrhage (PPH), obstetric anal sphincter injuries (OASIS).
Adverse neonatal outcome | Up to 48 hours postpartum
  stillbirth, infectious disease (sepsis, meningitis, pneumonia), 5-minute Apgar score < 7, umbilical artery pH < 7.0, NICU admission, RDS, use of mechanical ventilation, NEC.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Bachar, MD, Principal Investigator — Rambam Medical Health Center
Locations (1):
- Rambam, Ramat Yishai, Israel

IPD SHARING:
Plan to Share IPD: No